CLINICAL TRIAL: NCT06462885
Title: Living Alone is Predictive of Non-home Discharge Following Elective Total Hip Arthroplasty: a Matched-pairs Cohort Analysis
Status: Completed | Type: Observational
Sponsor: University of Virginia (Other)
Responsible Party: Principal Investigator, Zhiyi Zuo, MD, Principal Investigator, University of Virginia
Other Study IDs: HSRZOKZZ3
Record Dates: First submitted 2024-06-11; First posted 2024-06-17 (Actual); Last update posted 2024-06-18 (Actual); Status verified 2024-06

CONDITIONS: Arthropathy of Hip; Perioperative/Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Living alone: 1,624 patients undergoing elective total hip arthroplasty who were living alone at the time of admission.
  Interventions: Behavioral: home support, hiving alone
- Living with others: 1,624 patients undergoing elective total hip arthroplasty who were living with others at the time of admission.
  Interventions: Behavioral: home support, living with others

INTERVENTIONS:
Behavioral: home support, hiving alone — Home support: living alone
  Groups: Living alone
Behavioral: home support, living with others — Home support: living with others
  Groups: Living with others

SUMMARY:
The goal of this observational study is to assess the effect of living alone on total hip arthroplasty thirty-day outcomes. The main questions it aims to answer are:

Is living alone associated with discharge disposition (home versus non-home)? Is living alone associated with greater incidences of secondary adverse events?

Participants will be sampled from the 2021 American College of Surgeons National Surgical Quality Improvement Program

ELIGIBILITY:
Inclusion Criteria:

* Elective, non-emergent cases
* Living alone
* Living with others

Exclusion Criteria:

* Fracture in surgical diagnosis
* Hospital admission >1 day preoperatively
* End-stage renal disease (preoperative)
* Metastatic disease (preoperative)
* Sepsis (preoperative)
* Bleeding diathesis (preoperative)
* American Society of Anesthesiologists Physical Status Classification 5

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Elective total hip arthroplasty patients, ACS-NSQIP 2021
Sampling Method: Non-Probability Sample
Enrollment: 5677 (Actual)
Dates: Start 2021-01-01 (Actual); Primary Completion 2022-01-30 (Actual); Study Completion 2022-01-30 (Actual)

PRIMARY OUTCOMES:
Discharge disposition | Thirty days
  Home versus non-home

SECONDARY OUTCOMES:
Requiring home services | Thirty days
Functional status at discharge | Thirty days
  Dependent versus independent
Postoperative delirium | Thirty days
Hospital length of stay | Thirty days
Unplanned resource utilization | Thirty days
  Unplanned readmission and return to the operating room
Wound complications | Thirty days
  Superficial surgical site infection (SSI), deep incisional SSI, organ space SSI, and wound dehiscence
Systemic complications | Thirty days
  Cardiac arrest, myocardial infarction, stroke, reintubation, pneumonia, deep venous thrombosis, pulmonary embolism, bleeding, sepsis, septic shock, and acute kidney injury
Bleeding events | Thirty days
  Requiring transfusion
Mortality | Thirty days

CONTACTS AND LOCATIONS:
Overall Officials: Zhiyi Zuo, MD, PhD, Principal Investigator — University of Virginia
Locations (1):
- University of Virginia, Charlottesville, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
American College of Surgeons National Surgical Quality Improvement Program and the hospitals participating in the ACS NSQIP are the source of the data used herein. The Participant Use Data File (PUF) is a Health Insurance Portability and Accountability Act (HIPAA)-compliant data file containing cases submitted to the American College of Surgeons National Surgical Quality Improvement Program®. To request a copy of the PUF, individuals (data recipients) must agree to comply with the terms and conditions set forth in the Data Use Agreement, provide contact information, and complete a short online questionnaire. Once the information provided by the data recipient is received and processed by ACS NSQIP staff, a website address will be submitted electronically to the data recipient. The data recipient will then have 10 days (240 hours) to visit the website and download the data file.

REFERENCES:
- Available data/document: Individual Participant Data Set — https://www.facs.org/quality-programs/data-and-registries/acs-nsqip/participant-use-data-file/